CLINICAL TRIAL: NCT01786980
Title: The Methylation Phenotype Screening and Determination Mode Study of Liver Cancer Prognosis Related Gene
Status: Completed | Type: Observational
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, Department of Hepatic Surgery Ⅳ, Eastern Hepatobiliary Surgery Hospital
Other Study IDs: 2012ZX1000201600104
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma;; Radical Hepatic Resection;
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- liver cancer, Radical hepatic resection

SUMMARY:
Recurrence and metastasis are the main factors affecting the prognosis of liver cancer after curative resection. Establishing an effective prognostic evaluation method is able to not only assess patients' prognosis but also guide the treatment. At the same time, it helps us to gain knowledge of the mechanism underlying recurrence and metastasis of liver cancer and to provide the basis for the search for new effective intervention method.

In order to establish an effective prognostic evaluation method, we select liver cancer patients undergoing curative resection in our hospital. We plan to employ various technologies such as gene chip, methylation chip and flow cytometry to carry out comprehensive researches on liver cancer cell genetics, epigenetics, stem cells and tumor microenvironment changes. By analyzing clinical information including pathological features, patients' response to treatment, relapse, metastasis and survival, we aim to obtain the important factors affecting liver cancer prognosis, survival, recurrence and metastasis in order to be able to find and establish the effective prognostic evaluation method.

DETAILED DESCRIPTION:
Recurrence and metastasis are the main factors affecting the prognosis of liver cancer after curative resection. Establishing an effective prognostic evaluation method is able to not only assess patients' prognosis but also guide the treatment. At the same time, it helps us to gain knowledge of the mechanism underlying recurrence and metastasis of liver cancer and to provide the basis for the search for new effective intervention method.

In order to establish an effective prognostic evaluation method, we select liver cancer patients undergoing curative resection in our hospital. We plan to employ various technologies such as gene chip, methylation chip and flow cytometry to carry out comprehensive researches on liver cancer cell genetics, epigenetics, stem cells and tumor microenvironment changes. By analyzing clinical information including pathological features, patients' response to treatment, relapse, metastasis and survival, we aim to obtain the important factors affecting liver cancer prognosis, survival, recurrence and metastasis in order to be able to find and establish the effective prognostic evaluation method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with radical hepatectomy in Eastern Hepatobiliary Surgery Hospital;
2. Hepatocellular carcinoma confirmed pathologically;
3. The liver function is Child-Pugh A, as well as the Child-Pugh B achieved to A after treatment;
4. The HAI score of cirrhosis <12

Exclusion Criteria:

1. Patients with apparent cardiac, pulmonary, cerebric and renal dysfunction,which may affect the treatment of liver cancer.
2. Patients with other diseases which may affect the treatment mentioned here.
3. Patients with medical history of other malignant tumors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with radical hepatectomy in Eastern Hepatobiliary Surgery Hospital, and were confirmed hepatocellular carcinoma pathologically. The liver function was Child-Pugh A, as well as the Child-Pugh B achieved to A after treatment, and the HAI score of cirrhosis was <12.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2015

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality